CLINICAL TRIAL: NCT01431820
Title: Safety and Efficacy of Luliconazole Solution, 10% With Two Dosing Regimens in Distal Subungual Onychomycosis of the Toenails: A Randomized, Double-Blind, Vehicle-Controlled, Phase 2B/3 Study
Brief Title: Safety and Efficacy of Luliconazole Solution, 10% in Subjects With Mild to Moderate Onychomycosis
Acronym: SOLUTION
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Topica Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TP-1009-S; NCT01428856 (obsolete NCT alias)
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Distal and Lateral Subungual Onychomycosis
Keywords: Onychomycosis; Toenail Fungus; luliconazole; Antifungal; Topical
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Luliconazole Solution, 10% Regimen 1 (Experimental)
  Interventions: Drug: Luliconazole Solution, 10%
- Luliconazole Solution, 10% Regimen 2 (Experimental)
  Interventions: Drug: Luliconazole Solution, 10%
- Vehicle Solution Regimen 1 (Placebo Comparator)
  Interventions: Drug: Vehicle Solution
- Vehicle Solution Regimen 2 (Placebo Comparator)
  Interventions: Drug: Vehicle Solution

INTERVENTIONS:
Drug: Luliconazole Solution, 10% — Topical
  Arms: Luliconazole Solution, 10% Regimen 1; Luliconazole Solution, 10% Regimen 2
Drug: Vehicle Solution — Topical
  Arms: Vehicle Solution Regimen 1; Vehicle Solution Regimen 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a topical antifungal formulation, Luliconazole Solution, 10%, in the treatment of adults with onychomycosis of the toenails.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender, any race and between the ages of 18 and 70 inclusive
* Subjects with a clinical diagnosis with culture confirmation of distal subungual onychomycosis (DSO) - Subjects must be free of any disease that in the Investigator's opinion might interfere with the study evaluations or jeopardize the subject's safety

Exclusion Criteria:

* Subjects with a history of intolerance or hypersensitivity to imidazole compounds or the inactive components of the solution
* Subjects who are currently participating or have recently participated in another investigational medication or device study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who achieve complete cure of the target great toenail | Week 52

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Phoenix, Arizona
  - Los Angeles, California
  - San Diego, California
  - Denver, Colorado
  - Aventura, Florida
  - Miami, Florida
  - Boise, Idaho
  - Evansville, Indiana
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Detroit, Michigan
  - Fridley, Minnesota
  - Albuquerque, New Mexico
  - East Setauket, New York
  - Rochester, New York
  - Cincinnati, Ohio
  - Portland, Oregon
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - College Station, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Lynchburg, Virginia
  - Madison, Wisconsin

REFERENCES:
- See also: Safety and Tolerability of Luliconazole Solution, 10% in Patients with Moderate to Severe Distal Subungual Onychomycosis. Jones T, Tavakkol A. Antimicrob Agents Chemother. 2013 Apr 1. [Epub ahead of print] — http://www.ncbi.nlm.nih.gov/pubmed/23545529